CLINICAL TRIAL: NCT06475508
Title: Double-blind Multicenter Randomized Study of the Effectiveness and Safety of Tocilizumab Biosimilar (Complarate®) and Actemra® in Parallel Groups in Patients With Rheumatoid Arthritis With Repeated Intravenous Administration
Brief Title: Comparison of Complarate® (Tocilizumab Biosimilar) and Actemra® in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TZS-RA-III
Record Dates: First submitted 2024-06-20; First posted 2024-06-26 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Rheumatoid Arthritis
Keywords: tocilizumab; humanized monoclonal antibodies; safety; rheumatoid arthritis; equivalence; biosimilar; American College of Rheumatology (ACR); DAS28; disease-modifying anti-rheumatic drugs (DMARDs); rheumatic autoimmune disease; European League Against Rheumatism (EULAR); immunogenicity; Clinical Disease Activity Index (CDAI); Simplified Disease Activity Index (SDAI)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Throughout the study neither the investigators nor the patients knew which drug was being administered until the end of the comparative treatment study period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Complarate® (JSC "GENERIUM", Russia) (Experimental): tocilizumab biosimilar
  Interventions: Biological: Complarate®
- Actemra® (F. Hoffmann-La Roche Ltd., Switzerland) (Active Comparator): tocilizumab
  Interventions: Biological: Actemra®

INTERVENTIONS:
Biological: Complarate® — The investigational drug Complarate® was administered as an intravenous infusion at a dose of 8 mg/kg once every 4 weeks for 24 weeks.
  Other Names: tocilizumab biosimilar; GNR-087
  Arms: Complarate® (JSC "GENERIUM", Russia)
Biological: Actemra® — The reference drug Actemra® was administered as an intravenous infusion at a dose of 8 mg/kg once every 4 weeks for 24 weeks.
  Other Names: tocilizumab
  Arms: Actemra® (F. Hoffmann-La Roche Ltd., Switzerland)

SUMMARY:
This is a randomized double-blind comparative parallel group study of the efficacy and safety of tocilizumab biosimilar Complarate® and Actemra® in the treatment of patients with rheumatoid arthritis with moderate to high disease activity. Participants received an intravenous dose of tocilizumab 8 mg/kg once 4 weeks. The time on study treatment was 24 weeks.

DETAILED DESCRIPTION:
Complarate® (INN: tocilizumab) is being developed as a biosimilar to the drug Actemra®, a concentrate for the preparation of a solution for infusion.

Tocilizumab is a recombinant humanized monoclonal antibody to the human interleukin-6 (IL-6) receptor from the immunoglobulin G1 (IgG1) subclass of immunoglobulins. Tocilizumab binds to and inhibits both soluble and membrane IL-6 receptors.

This III phase study is aimed to compare the effectiveness, safety and immunogenicity of Complarate® and Actemra®. The study included patients aged 18-75 years at the time of signing the informed consent form with a documented diagnosis of rheumatoid artritis, established according to the 2010 ACR/EULAR classification criteria, at least 6 months before screening, with moderate or high degree of disease activity and insufficient response to methotrexate monotherapy (preservation of moderate/high disease activity for at least 3 months) and/or poor tolerability of methotrexate (including the subcutaneous form of the drug) and/or insufficient response to or intolerance to other synthetic disease-modifying anti-inflammatory drugs (sDMARDs) with or without methotrexate inclusive, who meet all criteria for participation in the study. The study included a screening period and a treatment period. Allocation of patients to treatment groups was carried out by randomization in a ratio of 2:1 to the study drug (Complarate®) and comparator drug (Actemra®). 465 patients (310 to the study drug group and 155 to the comparator drug group) were randomized.

ELIGIBILITY:
Inclusion Criteria:

* Availability of written informed consent obtained from the patient before the start of any procedures related to the study.
* Men and women 18-75 years of age, inclusive, at the time of signing the informed consent form.
* Patients with a documented diagnosis of rheumatoid artritis (RA), established according to the 2010 ACR/EULAR classification criteria at least 6 months before screening, with moderate to high disease activity and an insufficient response to methotrexate monotherapy (maintaining moderate/high disease activity for at least 3 months) and/or poor tolerability of methotrexate (including the subcutaneous form of the drug) and/or insufficient response to or intolerance to other synthetic disease-modifying anti-inflammatory drugs (sDMARDs) in combination with methotrexate or without methotrexate.
* The number of swollen and/or painful joints is 6 or more.
* No changes in the dosage regimen of standard RA therapy with oral glucocorticosteroids and NSAIDs for ≥ 4 weeks before screening.
* No changes in the dosing regimen of standard RA sDMARD therapy for ≥ 4 weeks before screening.
* Agreement to adhere to adequate methods of contraception throughout the study and for 3 months after the end of tocilizumab therapy.

Exclusion Criteria:

* A history of rheumatic autoimmune disease other than rheumatoid arthritis.
* Functional Class IV according to the ACR Functional Status Classification or wheelchair/bedridden.
* Development of pronounced extra-articular (systemic) manifestations of the disease and complications (rheumatoid vasculitis, amyloidosis, Felty's syndrome, neuropathy, damage to the organ of vision).
* Use of oral corticosteroids in doses greater than >10 mg daily prednisolone equivalent, or change in oral corticosteroid dose within 4 weeks before or during screening.
* Use of injectable corticosteroids (including intra-articular corticosteroids) or intra-articular hyaluronic acid injections within 4 weeks before or during screening.
* Therapy with tumor necrosis factor-alfa (TNF-alpha) inhibitors or any other genetically engineered biological drugs within 1 month before screening.
* History of tocilizumab therapy.
* Major surgery (including joint surgery) within 8 weeks before the start of the study or elective surgery within 6 months after the start of the study.
* A history of an adverse drug reaction to any of the components of the study drug or a reference drug.
* Immunization with any live or live attenuated vaccine within 1 month before the first dose of the study or comparator drug.
* A history of a disease associated with the accumulation of immune complexes (including serum sickness).
* Concomitant diseases and conditions that, in the opinion of the Investigator and/or Sponsor, jeopardize the safety of the patient during participation in the study, or which will influence the analysis of safety data.
* Active systemic infection (bacterial, viral or fungal) within 14 days before signing the informed consent form or at the time of screening.
* Blood donation or blood loss (450 ml of blood or more) less than 2 months before the start of the study.
* Pregnancy or breastfeeding.
* History of demyelinating disease of the central nervous system.
* History of diverticulosis/intestinal diverticulitis or chronic ulcerative diseases of the lower gastrointestinal tract, such as Crohn's disease, ulcerative colitis.
* History of tuberculosis.
* Positive/doubtful test with tuberculosis allergen.
* Participation in clinical trials of drugs less than 3 months before signing the informed consent form.
* Positive tests for hepatitis B or C, HIV or syphilis.
* Unwillingness or inability to comply with the recommendations prescribed by this protocol.
* Identification during screening of other diseases/conditions not listed above that, in the opinion of the physician-researcher, prevent the inclusion of the patient in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants with an American College of Rheumatology 20% (ACR20) response | week 24
  The ACR 20 response: greater than or equal to (>/=) 20 percent (%) improvement in TJC and SJC (28 assessed joints), and 20% improvement in 3 of the following 5 criteria, respectively: 1) PGDA, 2) PtGDA, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) CRP or ESR at week 24

SECONDARY OUTCOMES:
Proportion of Participants with an American College of Rheumatology 20% (ACR20), 50% (ACR50), and 70% (ACR70) Response | week 24
  The ACR 20, 50, and 70 responses: greater than or equal to (>/=) 20 percent (%), 50%, and 70% improvement in TJC and SJC (28 assessed joints), and 20%, 50%, 70% improvement in 3 of the following 5 criteria, respectively: 1) PGDA, 2) PtGDA, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) CRP or ESR at each visit
Time to ACR20 response | week 24
  The ACR 20 response: greater than or equal to (>/=) 20 percent (%) improvement in TJC and SJC (28 assessed joints), and 20% improvement in 3 of the following 5 criteria, respectively: 1) PGDA, 2) PtGDA, 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) CRP or ESR at week 24
Change in Disease Activity Score Based on 28-Joints Count (DAS28) | week 24
  DAS28 is calculated from the TJC and SJC based on a 28-joint assessment, the erythrocyte sedimentation rate (ESR) in millimeters per hour (mm/hour) and PtGDA assessed on 0-10 cm VAS. Higher scores indicate greater affectation due to disease activity. DAS28-ESR total score= 0-9.4. DAS28-ESR </=3.2 indicates low disease activity, DAS28-ESR >3.2 to 5.1 indicates moderate to high disease activity, and DAS28-ESR </=3.2 indicates remission.
Proportion of Participants With European League Against Rheumatism (EULAR) Response Based on DAS28 | week 24
  The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 </=3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to </=5.1 or change from baseline >0.6 to </=1.2 with DAS28 </=5.1; non-responders: change from baseline </=0.6 or change from baseline >0.6 and </=1.2 with DAS28 >5.1
Area under the curve (AUC) of the disease activity index (DAS28) | week 24
  DAS28 is calculated from the TJC and SJC based on a 28-joint assessment, the erythrocyte sedimentation rate (ESR) in millimeters per hour (mm/hour) and PtGDA assessed on 0-10 cm VAS. Higher scores indicate greater affectation due to disease activity. DAS28-ESR total score= 0-9.4. DAS28-ESR </=3.2 indicates low disease activity, DAS28-ESR >3.2 to 5.1 indicates moderate to high disease activity, and DAS28-ESR </=3.2 indicates remission.
Change in Simplified Disease Activity Index (SDAI) | week 24
  SDAI is a numerical sum of five outcome parameters: TJC and SJC based on a 28-joint assessment, PtGDA and PGDA assessed on 0-10 cm VAS and C-reactive protein (CRP) in milligrams per deciliter (mg/dL). Higher scores indicate greater affectation due to disease activity. SDAI total score = 0-86. SDAI </=3.3 indicates disease remission, >3.4 to 11 indicates low disease activity, >11 to 26 indicates moderate disease activity, and >26 indicates high disease activity
Change in Clinical Disease Activity Index (CDAI) | week 24
  CDAI is a numerical sum of 4 outcome parameters: tender joint count (TJC) and swollen joint count (SJC) based on a 28-joint assessment, patient's global assessment of disease activity (PtGDA) and physician global assessment of disease activity (PGDA) assessed on 0-10 centimeters (cm) visual analogue scale (VAS). Higher scores represent greater affectation due to disease activity. CDAI total score = 0-76. CDAI score less than or equal to (</=) 2.8 indicates disease remission, greater than (>) 2.8 to 10 indicates low disease activity, >10 to 22 indicates moderate disease activity, and >22 indicates high disease activity
Proportion of Participants who achieved remission in accordance with the ACR remission criteria | week 24
  Criteria for rheumatoid artritis remission (ACR/EULAR criteria, 2011). Simultaneous fulfillment of all conditions No. 1-4: 1. number of painful joints (TJ) ≤1, 2. number of swollen joints (SJ) ≤1, 3. C-reactive protein ≤1 mg/dL, 4. general assessment of the disease by the patient (OZB, according to YOUR) ≤1, OR fulfillment of condition No. 5, regardless of the fulfillment of conditions No. 1-4: 5. SDAI index ≤ 3.3.
Proportion of Participants who dropped out of the study due to insufficient treatment effectiveness | week 24
  Insufficient of therapy assessed as the lack of effect after 3 months of therapy using the disease activity in rheumatoid arthritis scale (DAS28) index (from less than 2.6 scores in remission to more then 5,1 scores for very active disease)

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — JSC GENERIUM
Locations (28):
- Russia (28):
  - Limited Liability Company "Family Clinic No. 4", Korolyov, Moscow Oblast
  - Limited Liability Company Research Medical Complex "Your Health", Kazan', Tatarstan Republic
  - State health care institution city clinical hospital №25, Volgograd, Volgograd Oblast
  - State Budgetary Healthcare Institution Chelyabinsk area Clinical Hospital, Chelyabinsk
  - Limited Liability Company "Medical Center "Revma-Med", Kemerovo
  - Limited Liability Company "OLLA-MED", Moscow
  - State Budgetary Healthcare Institution MKSC named after A.S. Loginova Moscow Health Department, Moscow
  - Federal State Budgetary Institution "Research Institute of Rheumatology named after V.A. Nasonova", Moscow
  - Federal State Autonomous Educational Institution of Higher Education First Moscow State Medical University named after I.M. Sechenov Ministry of Health of Russia, Moscow
  - Federal State Budgetary Educational Institution of Higher Education Moscow State University of Medicine and Dentistry, Moscow
  - Federal State Autonomous Educational Institution of Russian National Research Medical University named after. N. I. Pirogova, Moscow
  - Limited Liability Company "Ersi Medical", Novosibirsk
  - Limited Liability Company "Medical Center "Healthy Family", Novosibirsk
  - Federal State Budgetary Educational Institution of Higher Education Orenburg State Medical University of the Ministry of Health of Russia, Orenburg
  - Medical center, clinic "Medical Technologies", Saint Petersburg
  - Limited Liability Company "Ex Seven Clinical Research", Saint Petersburg
  - Limited Liability Company "Interleukin", Saint Petersburg
  - Limited Liability Company "Strategic Medical Systems", Saint Petersburg
  - State Budgetary Healthcare Institution Leningrad area Clinical Hospital, Saint Petersburg
  - JSC "North-West Center for Evidence-Based Medicine", Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education Saratov State Medical University named after. V.I.Razumovsky Ministry of Health of Russia, Saratov
  - Private foundation "RZD-Medicine" Smolensk", Smolensk
  - State Budgetary Healthcare Institution Tula area Clinical Hospital, Tula
  - State Budgetary Healthcare Institution Ulyanovsk area Clinical Hospital, Ulyanovsk
  - Limited Liability Company "CMKI-PRACTIKA", Yaroslavl
  - State Budgetary Healthcare Institution "Clinical Hospital No. 2", Yaroslavl
  - Central City Hospital, Yaroslavl
  - JSC "TsSM", Yekaterinburg

IPD SHARING:
Plan to Share IPD: No